CLINICAL TRIAL: NCT00294125
Title: Flavocoxid: A Medical Food Therapy for Osteoarthritis
Brief Title: Flavocoxid, A Plant-Derived Therapy, for the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Primus Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sarah Morgan, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R41AR051232 (NIH); R41AR051232 (NIH); 1R41AR051232-01A1 (NIH)
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Osteoarthritis
Keywords: Medical Food; Botanicals; Phytochemicals
MeSH Terms: conditions — Osteoarthritis | interventions — flavocoxid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Participants will receive daily flavocoxid for 12 weeks.
  Interventions: Drug: Flavocoxid
- 2 (Placebo Comparator): Participants will receive placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flavocoxid — Daily flavocoxid for 12 weeks
  Arms: 1
Drug: Placebo — Daily placebo for 12 weeks
  Arms: 2

SUMMARY:
Nonsteroidal anti-inflammatory drugs (NSAIDs) are commonly prescribed to treat arthritis. The purpose of this study is to test the effectiveness of flavocoxid, a plant-derived compound, for the treatment of knee osteoarthritis (OA) in adults.

Study hypotheses: 1) Flavocoxid has an acceptable safety and tolerability profile as determined by the Generally Regarded as Safe (GRAS) profile in patients with OA compared to identical placebo. 2) Flavocoxid will be more effective as a therapy for OA compared to identical placebo.

DETAILED DESCRIPTION:
OA is a leading chronic disease in older adults and is characterized by degeneration of articular cartilage of the joints in hands, spine, knees, and hips. In joints, tissue injury and pain are caused by the conversion of arachidonic acid to such inflammatory compounds as cyclooxygenases-1 and -2 (COX-1 and -2) and 5-lipoxygenase (5-LO). Conventional NSAIDs inhibit COX-1 and -2, but have little or no effect on 5-LO. NSAIDs provide relief from the pain of OA; however, NSAIDS are also associated with significant side effects, including gastrointestinal bleeding, venous thrombosis, and nephrotoxicity. Novel alternative therapies with increased safety and efficacy with fewer or no side effects are desirable; plant-derived substances might be useful alternatives to NSAIDs. Flavocoxid, a botanical extract derived from two plants, Scutellaria baicalensis and Acacia catechu, has been shown to inhibit COX-1 and -2 as well as 5-LO. The purpose of this study is to evaluate the safety and efficacy of flavocoxid in relieving the symptoms of knee OA in adults.

This study will last 12 weeks. Participants will be randomly assigned to one of two groups. Group 1 participants will receive daily flavocoxid; Group 2 participants will receive placebo. There will be 5 study visits: study entry and Weeks 2, 4, 8, and 12. Joint pain, tenderness, and swelling will be assessed at each study visit. A 30-foot timed walking test will also be performed at all visits. A physical exam and blood collection will occur at study entry and Week 12. Other study assessments will include safety monitoring, patient/physician global disease ratings, quality of life measures, depression and anxiety ratings, and measures of efficacy as determined by the Western Ontario and McMaster (WOMAC) OA index.

ELIGIBILITY:
Inclusion Criteria:

* Meet American College of Rheumatology (ACR) clinical criteria for knee OA
* In good medical and psychological health
* Able and willing to discontinue NSAIDs, natural therapies, and other pain medications for OA for 1 week prior to the first study visit and also throughout the course of the clinical trial
* Knee pain rated greater than 4 cm on a 10 cm visual analog scale (VAS)
* Intends to stay in the area and complete the 12-week protocol
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Serious or unstable concomitant medical or psychological illnesses that would impair the patient's ability to complete the study
* Significant cardiac disease OR history of myocardial infarction in the 12 months prior to study entry
* Uncontrolled hypertension
* Significant bleeding disorders. Participants who have bleeding disorders related to uncontrolled, bleeding hemorrhoids occurring in the 12 months prior to study entry are not excluded.
* Uncontrolled gastrointestinal disease resulting in bleeding in the 60 days prior to study entry. Participants with controlled and uncomplicated ulcers are not excluded.
* Inflammatory arthritis, gout, pseudogout, Paget's disease, or any chronic pain syndrome
* Severe pes anserine bursitis, acute joint trauma, or complete loss of articular cartilage on the index knee
* Intravenous, intramuscular, or intra-articular steroids to the index joint within 60 days of study screening
* Alcohol, intravenous drug, or prescription drug abuse
* Investigational drugs within 30 days of study screening
* Current use of anticoagulants such as warfarin
* Oral corticosteroids or other immunosuppressants within 6 months of study screening
* Severe psoriasis requiring use of biologic immunomodulators such as alefacept, etanercept, infliximab, or cyclosporine
* Hypersensitivity to analgesics, cyclo-oxygenase inhibitors, lipoxygenase inhibitors, or flavonoids
* Pregnancy or breastfeeding

Exclusion Criteria Postenrollment:

* Abnormal laboratory test results at study screening, as determined by the investigator
* Liver enzyme levels (SGOT, SGPT, alkaline phsphatase) two times the upper limit of normal
* Leukocyte counts less than 3.5 times 109/L or platelet counts less than 150 times 109/L
* At increased risk for cardiovascular problems based on the Framingham Cardiac Risk assessment questionnaire
* Kellgren/Lawrence radiographic score of 0, 1, or 4 on x-ray of index joint taken within 12 months of study entry
* Impaired renal function (creatinine greater than 1.5 mg/dl)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of flavocoxid (clinical status; causality and occurrence of adverse events) | Measured throughout 12-week treatment period

SECONDARY OUTCOMES:
Efficacy of treatment and clinical benefit | Measured at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L. Morgan, MD, RD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Morgan SL, Baggott JE, Moreland L, Desmond R, Kendrach AC. The safety of flavocoxid, a medical food, in the dietary management of knee osteoarthritis. J Med Food. 2009 Oct;12(5):1143-8. doi: 10.1089/jmf.2008.0244. PMID 19857081